CLINICAL TRIAL: NCT02666859
Title: The Use of Virtual Reality to Enhance Upper Limb Prosthetic Training and Rehabilitation
Brief Title: Virtual Reality Prosthetic Training and Rehabilitation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Telemedicine & Advanced Technology Research Center (Other)
Responsible Party: Principal Investigator, Stephanie L. Carey, Research Coordinator, University of South Florida
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00016934
Record Dates: First submitted 2016-01-12; First posted 2016-01-28 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Amputation of Upper Limb

STUDY DESIGN:
Intervention Model Description: Virtual Reality Prosthetic Training
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unilateral Transradial Amputation (Experimental): This group includes people with a unilateral transradial amputation. Potential subjects must use a body-powered or myoelectric prosthetic device. This group will be exposed to virtual reality therapy and non-virtual reality therapy.
  Interventions: Device: Virtual Reality
- Unilateral Transhumeral Amputation (Experimental): This group includes people with a unilateral transhumeral amputation. Potential subjects must use a body-powered or myoelectric prosthetic device. This group will be exposed to virtual reality therapy and non-virtual reality therapy.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — During this intervention, the subjects will be immersed in a virtual reality system called the Computer Assisted Rehabilitation Environment (CAREN) system to complete the tasks.

SUMMARY:
The proposed project is to develop an effective prosthetic training and rehabilitation regimen, with the use of virtual reality, to return patients to the highest level of independence and functioning possible. The Computer Assisted Rehabilitation Environment (CAREN) system (Motek Medical, Netherlands) will be used to immerse patients into real life situations while providing real time visual feedback of their motion to improve the training and rehabilitation of upper limb prosthetic users.

DETAILED DESCRIPTION:
The subjects will be asked to participate in two 1-2 hour sessions to test the range of motion (ROM), activities of daily living ( ADL) and return to duty tasks (RTD) tasks with and without the use of virtual reality. All amputee subjects will be required to wear their same preferred prosthetic device for all sessions. The ROM tasks include, elbow flexion/extension, forearm pronation/supination, shoulder flexion/extension, shoulder abduction/adduction, shoulder rotation, torso flexion/extension, torso lateral flexion, and torso rotation. The ADL tasks would include a series of tasks to encompass typical actives one would encounter on a daily basis such as, drinking from a cup, bilateral and unilateral lift tasks, and a reach and grasp test. The RTD tasks would include a series of simple tasks service members typically perform in their daily work routine such as donning and doffing a jacket and helmet, packing and unpacking a rucksack, and carrying a weapon.

The subjects will be asked to complete each task three times. Prior to performing a task, when participating in the virtual reality session, the task will be demonstrated on the virtual screen with an animated model. The motion of the animated model will be determined by previously collected data to accurately predict the correct motion for each individual. An avatar of the subject will then be shown on the screen to display the real time motion. The reflective markers that were strategically placed on the subject will be connected to the corresponding joint on the virtual avatar to accurately animate the real time motion of the subject on the virtual screen. The demonstrated model will be shown simultaneously with the real time avatar to show the accuracy of the subject's performance in relation to the individualized predicted optimized motion. This will provide instant visual feedback to the subject.

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral transhumeral or transradial amputation
* uses body-powered or myoelectric prosthetic device.
* free of any health aliment that would impair physical function
* must not have any injuries or surgeries on the affected limb within the past 90 days.
* Subjects ,just be able to perform activities of daily living without assistance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Joint Angle Range of Motion | 2 hours
  Using a motion capture system, joint angle measurements will be taken throughout the sessions while the subject completes the tasks.

SECONDARY OUTCOMES:
Movement Symmetry | 2 hours
  Using a motion capture system and the joint angle measurements, the movement symmetry of the arms will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Knight, M.S. BME, Principal Investigator — University of South Florida; Stephanie Carey, Ph.D. BME, Study Director — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States